CLINICAL TRIAL: NCT07292441
Title: A Multicenter Extension Study of the Phase 3 Clinical Study of GZR18 Injection for Weight Loss
Brief Title: Extension Study of the Phase 3 Clinical Study of GZR18 Injection for Weight Loss
Acronym: GZR18-BWM-303
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZR18-BWM-303
Record Dates: First submitted 2025-11-20; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- GZR18 injection Dose1 (Experimental)
  Interventions: Drug: GZR18 injection
- GZR18 injection Dose2 (Experimental)
  Interventions: Drug: GZR18 injection
- GZR18 injection Dose3 (Experimental)
  Interventions: Drug: GZR18 injection

INTERVENTIONS:
Drug: GZR18 injection — Used as specified in the protocol
  Arms: GZR18 injection Dose1; GZR18 injection Dose2; GZR18 injection Dose3
Other: Placebo — Administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
This is a Phase 3 extension study conducted in subjects who have received GZR18 Injection once every 2 weeks (Q2W) for weight loss treatment for 52 weeks, aiming to explore the effect and safety of continuous injection of GZR18 Injection once every 4 weeks (Q4W) for 24 weeks on body weight.

In this study, it is planned to include subjects who have participated in the original study and completed the study contents of the original protocol. All subjects will maintain a regular diet and exercise lifestyle during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who participated in the original study, completed the last dose at W50, EOT visit at W52 and safety follow-up visit at W55 of either original study, with last dose at W50 ≥ 24 mg (including blinded dose of placebo).
2. Subjects with BMI > 18.5 kg/m² at W55 of the original study and before randomization at Visit 2 (V2) of this study, who are assessed by the investigator as suitable for participating in this study.
3. Subjects of childbearing potential with no birth plan from the signing of ICF to 8 weeks after the last dose, willingness to take effective contraceptive measures, and no plan for sperm or ovum donation. Non-lactating women of childbearing potential (WOCBP) with a negative pregnancy test result before randomization at V2 in this study.
4. Able to understand the procedures and methods of this study, willing and able to maintain a regular diet and exercise lifestyle during the study period, willing and able to undergo subcutaneous injections of the investigational medicinal product (IMP), and willing to sign the ICF voluntarily.

   -

Exclusion Criteria:

1. Subjects who used Semaglutide (Wegovy®) in the original study.
2. Subjects with a previous diagnosis of any type of diabetes mellitus (excluding gestational diabetes mellitus).
3. Subjects with FPG ≥ 7.0 mmol/L or HbA1c ≥ 6.5% in the central laboratory test at W52 visit of the original study.
4. Subjects who plan to participate in another clinical study of an investigational medicinal product or device, or receive drug or non-drug therapies that affect body weight (excluding diet and exercise control) before completing all scheduled assessments in this clinical study.
5. Subjects with any other factors (including but not limited to previous compliance in the original study) that may affect the efficacy or safety evaluation of this study as judged by the investigator.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percent change (%) from baseline in body weight | from Week 0 (W0) to Week 24 (W24)

SECONDARY OUTCOMES:
Changes from baseline in weight; | from Week 0 (W0) to Week 24 (W24)
Changes from baseline body mass index (BMI)； | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in waist circumference, hip circumference, and waist-hip ratio (waist circumference/hip circumference)； | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in hemoglobin A1c (HbA1c) ; | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in fasting plasma glucose (FPG); | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in blood pressure (SBP and DBP); | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in total cholesterol (TC); | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in low-density lipoprotein cholesterol (LDL-C); | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in high-density lipoprotein cholesterol (HDL-C); | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in triglyceride (TG); | from Week 0 (W0) to Week 24 (W24)
Changes from baseline in free fatty acids. | from Week 0 (W0) to Week 24 (W24)
Treatment-Emergent Adverse Events (TEAEs); | from Week 0 (W0) to Week 25 (W25)
Treatment-Emergent Serious Adverse Events (TESAEs); | from Week 0 (W0) to Week 25 (W25)
Pulse rate; | from Week 0 (W0) to Week 25 (W25)
Lipase; | from Week 0 (W0) to Week 25 (W25)
Amylase; | from Week 0 (W0) to Week 25 (W25)
Calcitonin | from Week 0 (W0) to Week 25 (W25)
The scores of Patient Health Questionnaire-9 | from Week 0 (W0) to Week 25 (W25)
  the highest/worst score during the trial (the higher scores mean a worse outcome
GZR18 anti-drug antibody (ADA) and neutralizing antibody (NAb); | from Week 0 (W0) to Week 25 (W25)
Cross reaction between GZR18 ADA and endogenous glucagon-like peptide-1 (GLP-1). | from Week 0 (W0) to Week 25 (W25)

CONTACTS AND LOCATIONS:
Locations (1):
- Study site 01, Beijing, Beijing Municipality, China